CLINICAL TRIAL: NCT06661330
Title: Exploring Gender Differences in the Effects of Diet and Physical Activity on Metabolic Parameters
Acronym: GENDIET
Status: Completed | Type: Observational
Sponsor: San Raffaele Telematic University (Other)
Responsible Party: Principal Investigator, Mauro Lombardo, Associate professor, San Raffaele Telematic University
Other Study IDs: Gender_Diet_2024
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Diet Therapy; Mediterranean Diet; Body Composition Changes; Physical Activity
Keywords: Metabolic parameters; Mediterranean diet; Physical activity; Body composition; Lipid profiles; Gender differences
MeSH Terms: conditions — Motor Activity | interventions — Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mediterranean Diet Intervention Group: This group consists of 200 adults who participated in a 6-month Mediterranean diet intervention combined with regular physical activity. The intervention focused on reducing energy intake by approximately 600 kcal/day while emphasizing plant-based foods, fish, and poultry. Participants' metabolic parameters, including body composition, fasting glucose, lipid profiles, and liver enzymes, were assessed at baseline and after 6 months.
  Interventions: Other: Behavioral Treatment

INTERVENTIONS:
Other: Behavioral Treatment — Participants followed a 6-month hypocaloric Mediterranean-style diet, reducing energy intake by approximately 600 kcal/day. The diet emphasized fruits, vegetables, whole grains, and fish, while limiting red meat and processed foods. Additionally, participants were required to perform moderate physical activity, including 50 minutes of aerobic exercise, 3 times a wee

SUMMARY:
This study investigates the gender-specific effects of diet and physical activity on metabolic parameters in a cohort of adults. The study involved a 6-month intervention based on a Mediterranean-style diet and regular physical activity, with the primary objective of assessing changes in body composition, fasting glucose, lipid profiles, and liver enzymes. Participants were stratified by gender to evaluate whether men and women exhibit different metabolic responses to the intervention. The results aim to provide insights into personalized nutritional recommendations based on gender differences.

DETAILED DESCRIPTION:
The study was conducted to explore gender differences in metabolic responses to a Mediterranean-style diet combined with a structured physical activity regimen. The study population included 2,509 participants recruited from a metabolic health clinic in Rome, Italy. Participants followed a 6-month hypocaloric diet, with macronutrient distribution of 16% protein, 25% fats, and 59% carbohydrates. The diet emphasized plant-based foods, with limited red meat consumption and regular intake of fish and poultry. Alongside the dietary intervention, participants were instructed to perform moderate physical activity, including aerobic exercises for 50 minutes, three times a week.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Able to follow a Mediterranean diet and participate in physical activity.
* Provide informed consent.

Exclusion Criteria:

* Pregnant women.
* Individuals with severe chronic diseases.
* Participants with alcohol or substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes 200 adults from a metabolic health clinic in Rome, Italy, participating in a 6-month Mediterranean diet and physical activity intervention.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Composition (Fat Mass and Lean Mass) | Baseline and 6 months
  The primary outcome is the change in body composition, specifically fat mass and lean mass, after a 6-month Mediterranean diet intervention combined with regular physical activity.

SECONDARY OUTCOMES:
Change in Fasting Glucose | Baseline and 6 months
  The secondary outcome includes changes in fasting glucose measured at baseline and after the 6-month intervention.
Change in Lipid Profiles (HDL, LDL, Total Cholesterol, Triglycerides) | Baseline and 6 months
  The secondary outcome includes changes in lipid profiles (HDL, LDL, total cholesterol, and triglycerides) measured at baseline and after the 6-month intervention.
Change in Creatinine Levels | Baseline and 6 months
  The secondary outcome includes changes in creatinine levels measured at baseline and after the 6-month intervention.
Change in Liver Enzymes (AST, ALT) | Baseline and 6 months
  The secondary outcome includes changes in liver enzymes (AST, ALT) measured at baseline and after the 6-month intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Caprio, PhD, Study Director — Department for the Promotion of Human Science and Quality of Life San Raffaele Open University, Rome
Locations (1):
- Department for the Promotion of Human Science and Quality of Life San Raffaele Open University, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The de-identified individual participant data (IPD) will be made available to researchers upon reasonable request. Data will be shared securely for the purpose of secondary research.

REFERENCES:
- [Background] Manzano-Carrasco S, Felipe JL, Sanchez-Sanchez J, Hernandez-Martin A, Clavel I, Gallardo L, Garcia-Unanue J. Relationship between Adherence to the Mediterranean Diet and Body Composition with Physical Fitness Parameters in a Young Active Population. Int J Environ Res Public Health. 2020 May 11;17(9):3337. doi: 10.3390/ijerph17093337. PMID 32403376
- [Background] Barrea L, Verde L, Suarez R, Frias-Toral E, Vasquez CA, Colao A, Savastano S, Muscogiuri G. Sex-differences in Mediterranean diet: a key piece to explain sex-related cardiovascular risk in obesity? A cross-sectional study. J Transl Med. 2024 Jan 10;22(1):44. doi: 10.1186/s12967-023-04814-z. PMID 38200498
- [Derived] Gorini S, Camajani E, Cava E, Feraco A, Armani A, Amoah I, Filardi T, Wu X, Strollo R, Caprio M, Padua E, Lombardo M. Gender differences in eating habits and sports preferences across age groups: a cross-sectional study. J Transl Med. 2025 Mar 12;23(1):312. doi: 10.1186/s12967-025-06311-x. PMID 40075461
- [Derived] Gorini S, Camajani E, Feraco A, Armani A, Karav S, Filardi T, Aulisa G, Cava E, Strollo R, Padua E, Caprio M, Lombardo M. Exploring Gender Differences in the Effects of Diet and Physical Activity on Metabolic Parameters. Nutrients. 2025 Jan 20;17(2):354. doi: 10.3390/nu17020354. PMID 39861484